CLINICAL TRIAL: NCT02395471
Title: Assessment of a Minimally Invasive Esophageal Cytology Collection System in Patients With Barrett's Esophagus or GERD Symptoms
Brief Title: Cytosponge Adequacy Study Evaluation II
Acronym: CASEII
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medtronic - MITG (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: B-271
Record Dates: First submitted 2015-03-12; First posted 2015-03-23 (Estimated); Results first posted 2019-07-30 (Actual); Last update posted 2019-07-30 (Actual); Status verified 2019-07

CONDITIONS: Barrett's Esophagus; GERD
MeSH Terms: conditions — Barrett Esophagus; Gastroesophageal Reflux

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Patient wth Barrett's (Experimental): Subjects presenting for routine endoscopic BE surveillance examinations
  Interventions: Device: Cytosponge™ Cell Collection Device
- Patients with GERD (Experimental): Subjects with gastroesophageal reflux disease (GERD) symptoms undergoing upper endoscopy for screening for BE
  Interventions: Device: Cytosponge™ Cell Collection Device

INTERVENTIONS:
Device: Cytosponge™ Cell Collection Device — Cytosponge™ Cell Collection Device is indicated for use in the collection and retrieval of surface cells in the esophagus.

SUMMARY:
This study will assess the Minimally Invasive Esophageal Cytology Collection System in Patients with Barrett's Esophagus or GERD Symptoms.

DETAILED DESCRIPTION:
This is a cross-sectional study of subjects with Barrett's esophagus (BE) to assess the utility of the Cytosponge device as a non-endoscopic method for collecting surface cells from the esophagus. This study will enroll 2 groups of subjects: 1) Subjects presenting for routine endoscopic BE surveillance examinations (n=120), and 2) Subjects with gastroesophageal reflux disease (GERD) symptoms undergoing upper endoscopy for screening for BE (n=55). After informed consent, and on the same day as the endoscopic procedure, the subject will undergo administration of the Cytosponge device and complete a questionnaire. The subject will then undergo routine upper endoscopy, with assessment of BE (where applicable), and biopsy per accepted surveillance or screening recommendations. The Cytosponge will be placed in fixative and shipped to an accredited pathology laboratory for embedding in paraffin and hematoxylin and eosin (H&E) staining to assess the adequacy of the specimen. Further evaluation of the specimen may be performed using trefoil factor 3 (TFF3). If the Cytosponge tissue specimen is inadequate, the subject will be recalled for a repeat sponge procedure (not endoscopy) 30 days later. Routine care tissue biopsies will undergo standard processing and H&E staining at the home institution, with assessment by expert gastrointestinal pathologists. Subjects will be contacted via phone 7 days (+/- 2 days) after Cytosponge administration to complete additional questionnaires and assess adverse events.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female subjects, age 18 and above.
2. Able to read, comprehend, and complete the consent form.
3. Clinically fit for an endoscopy.
4. a) Previous confirmed diagnosis of Barrett's esophagus with intestinal metaplasia, and Prague classification of at least one circumferential centimeter of BE or a total BE segment length of at least 3 centimeters (C1+ or CXM3+) (BE arm) . OR b) If the subject does not have documented Prague Classification prior to screening, but the PI is convinced that the subject will meet the inclusion criteria based on previous documentation (for instance, mention of "long-segment BE," they may enroll the subject in the study at their discretion. The study upper endoscopy must confirm that the subject has C1+ or CXM3+ (BE arm). If (C1+ or CXM3+) is not observed at the time of study endoscopy, the subject may still be enrolled but not included in the data analysis with the BE cohort. The data may be analyzed in a separate cohort. OR c) Self-reported heartburn or regurgitation on at least a monthly basis for at least 6 months (GERD arm).

Exclusion Criteria:

1. Individuals with a diagnosis of an oropharynx, esophageal or gastro-esophageal tumor, or symptoms of dysphagia.
2. Any history of esophageal varices, stricture, or prior dilation of the esophagus.
3. Current use of anti-thrombotics (anti-coagulants and anti-platelet drugs) that cannot be safely discontinued for the appropriate drug-specific interval in the peri-administration period. Depending on the particular agent or reason for the anti-thrombotic therapy, it may not be necessary to discontinue anti-thrombotic agents. There could be circumstances where the drug may not need to be discontinued if the risk of bleeding is considered negligible (e.g. daily aspirin therapy). Physicians should use their clinical judgement and should consult guidelines such as those provided by the ASGE.
4. Known bleeding disorder.
5. Individuals who have had a myocardial infarction or any cardiac event < 6 months prior to enrollment.
6. Individuals who have had a cerebrovascular event < 6 months prior to enrollment in which swallowing was affected.
7. Prior ablative or resection therapy of the esophagus including radiofrequency ablation (RFA), photodynamic therapy (PDT), spray cryotherapy, endoscopic mucosal resection, and other ablation therapies.
8. Any history of esophageal surgery, except for uncomplicated fundoplication.
9. Do not need upper endoscopy as part of patient management.
10. Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 191 (Actual)
Dates: Start 2015-08; Primary Completion 2018-04-24 (Actual); Study Completion 2018-06-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Amanda Cafaro, BSN, Study Director — Medtronic Clinical Research Director
Locations (5):
- United States (5):
  - Univeristy of California, Los Angeles, Los Angeles, California
  - University of Colorado, Aurora, Colorado
  - Northwestern University, Chicago, Illinois
  - University of North Carolina, Chapel Hill, North Carolina
  - Gastrointestinal Associates, Knoxville, Tennessee

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Patient Wth Barrett's | Patients With GERD
Started | 129 | 62
Completed | 122 | 59
Not Completed | 7 | 3
Not completed — Lost to Follow-up | 2 | 0
Not completed — Withdrawal by Subject | 2 | 1
Not completed — Physician Decision | 1 | 0
Not completed — Protocol Violation | 0 | 1
Not completed — Failure to swollow sponge twice | 1 | 0
Not completed — Patient did not return for procedure | 0 | 1
Not completed — Subject not eligible | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Patient Wth Barrett's | Patients With GERD | Total
Number analyzed (Participants) | 129 | 62 | 191
Age, Continuous [Mean (Standard Deviation); unit: years] | 64 (10.4) | 54.2 (15.1) | 60.8 (12.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 36 | 39 | 75
  Male | 93 | 23 | 116
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 4 | 6
  Not Hispanic or Latino | 127 | 57 | 184
  Unknown or Not Reported | 0 | 1 | 1
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — In Patients with GERD, one patient was both American Indian Or Alaska Native and Asian.
  Participants
    American Indian Or Alaska Native | 0 | 1 | 1
    Asian | 1 | 2 | 3
    Black or African American | 0 | 5 | 5
    Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
    White | 127 | 52 | 179
    Other | 1 | 2 | 3

OUTCOME MEASURES:

1. Primary Outcome: Procedure Preference and Acceptability Questionnaire and Visual Analog Scale
Description: The first primary objective of the study was to assess the acceptability of a novel, minimally invasive esophageal mucosal sampling technique, the Cytosponge™, in subjects undergoing surveillance of BE who have had at least a C1 or M3 segment confirmed, and 2) in subjects with GERD undergoing screening for BE. This includes measures of acceptability as demonstrated on the Impact of Event Scale, a Visual Analog Scale for Pain, and the subject's willingness to undergo repeat Cytosponge™ administration if it were offered to him/her. The Visual Analog Scale is measured from 0-100 scale for pain, 0 representing no pain and 100 representing the highest level of pain.
Time Frame: Immediately post procedure up to 7 days +/- 3 days
Measure: Mean (Standard Deviation); unit: Units on a scale
Groups:
- Study Participant Cytosponge Procedure Acceptability: Acceptability of the Cytosponge Procedure by all study subjects that underwent both Cytosponge and Endoscopy
Arm/Group | Study Participant Cytosponge Procedure Acceptability
Number analyzed (Participants) | 191
Units on a scale
  On scale of 0-10 (10-high), rate Cytosponge exper. | 7.2 (2.5)
  On scale of 0-10 (10-high), rate endoscopy exper. | 8.5 (2.5)
  Diff. between the two scales: (Cyto/Endoscop) | -1.3 (2.4)
  Visual Analog Scale | 16.2 (18.3)

2. Primary Outcome: Number of Participants With Adequate Cytosponge™ Sample
Description: To assess the adequacy of cytology samples obtained by Cytosponge in this population after 1 sampling, and after 2 samplings if first sample inadequate.
Time Frame: Immediately post procedure up to 7 days +/- 3 days
Measure: Count of Participants; unit: Participants
Arm/Group | Patient Wth Barrett's | Patients With GERD
Number analyzed (Participants) | 127 | 61
Participants | 115 | 56

3. Secondary Outcome: Operating Characteristics
Description: The operating characteristics of this technique against a gold standard of upper endoscopy with biopsies for endoscopic surveillance in subjects with BE who demonstrate an adequate sample on Cytosponge assessment.
Time Frame: Immediately post procedure up to 7 days +/- 3 days
Measure: Number (95% Confidence Interval); unit: Percentage
Groups:
- Operating Characteristics of Cytosponge™/TFF3 vs BE Diagnosis: Sensitivity, Specificity, PPV, NPV, and Accuracy of Cytosponge™/TFF3 vs. the Gold Standard of Endoscopy for BE Diagnosis
Arm/Group | Operating Characteristics of Cytosponge™/TFF3 vs BE Diagnosis
Number analyzed (Participants) | 154
Percentage
  Sensitivity | 75.5 [65.6 to 83.8]
  Specificity | 76.7 [64 to 86.6]
  Positive Predictive Value | 83.5 [73.9 to 90.7]
  Accuracy | 76 [68.4 to 82.5]

4. Secondary Outcome: Cytosponge™ Operating Characteristics vs Worst Histology Ever
Description: The second secondary objective was to assess the operating characteristics of Cytosponge™ against the worst ever histology documented in the subject.
Time Frame: Immediately post procedure up to 7 days +/- 3 days
Measure: Number (95% Confidence Interval); unit: Percentage
Groups:
- Cytosponge™ Operating Characteristics vs Worst Histology: The second secondary objective was to assess the operating characteristics of Cytosponge™ against the worst ever histology documented in the subject.
Arm/Group | Cytosponge™ Operating Characteristics vs Worst Histology
Number analyzed (Participants) | 158
Percentage
  Sensitivity | 77 [67.5 to 84.8]
  Specificity | 81 [68.6 to 90.1]
  Positive Predictive Value | 87.5 [78.7 to 93.6]
  Negative Predictive Value | 67.1 [54.9 to 77.9]
  Accuracy | 78.5 [71.2 to 84.6]

5. Secondary Outcome: Cytosponge™ Operating Characteristics as a Function of Baseline Histology
Description: The third secondary objective was to assess the operating characteristics of Cytosponge™ as a function of baseline histology. At the outset of this study, no data was available regarding the accuracy of TFF3 in samples collected by Cytosponge™ in subjects with BE and more advanced disease (low-grade dysplasia and high-grade dysplasia). These subjects are at greatest risk for progression to cancer. We planned to collect pilot data on operating characteristics of the assay by degree of baseline dysplasia. We hypothesized that TFF3 would perform with similar operating characteristics in this group compared to non-dysplastic BE.
Time Frame: Immediately post procedure up to 7 days +/- 3 days
Population: Among study subjects with BE that exhibited HGD, there were no true negatives or false positives, therefore specificity of the assay was not calculated for this subgroup.
Measure: Number; unit: Percentage
Groups:
- Non-Dysplastic BE: Non-Dysplastic BE
- Indefinite for Dysplasia: Indefinite for Dysplasia
- Low Grade Dysplasia: Low Grade Dysplasia
- High Grade Dysplasia: High Grade Dysplasia
Arm/Group | Non-Dysplastic BE | Indefinite for Dysplasia | Low Grade Dysplasia | High Grade Dysplasia
Number analyzed (Participants) | 77 | 13 | 10 | 6
Percentage
  Sensitivity | 76.2 | 66.7 | 77.8 | 83.3
  Specificity | 64.3 | 100 | 0 | NA — Analysis not available, See Population Description.
  Accuracy | 74.0 | 69.2 | 70.0 | 83.3

6. Secondary Outcome: Summary of Abrasion, Bleeding, and Perforation Observed Via Endoscopy
Description: The fourth secondary objective was to assess the degree of mucosal abrasion following Cytosponge™ administration, using a standardized scale. The incidence is presented in the data below for abrasion, bleeding and perforation observed during Endoscopy.
Time Frame: Immediately post procedure up to 7 days +/- 3 days
Measure: Count of Participants; unit: Participants
Groups:
- Incidence: Incidence of Abrasion, Bleeding and Perforation observed via Endoscopy
Arm/Group | Incidence
Number analyzed (Participants) | 190
Participants
  Abrasion | 117
  Bleeding | 58
  Bleeding-From Cytosponge contact site | 14
  Bleeding-From Biopsy Site | 56
  Perforation | 0
  Any of These 3 Conditions | 141

7. Secondary Outcome: Ongoing Safety Measures
Description: To collect and analyze ongoing safety measures of Cytosponge use in the target population.
Time Frame: Immediately post procedure up to 7 days +/- 3 days
Measure: Count of Participants; unit: Participants
Groups:
- Incidence of AE's: Incidence of AE's
Arm/Group | Incidence of AE's
Number analyzed (Participants) | 14
Participants
  Not Coded | 3
  Dyspepsia | 1
  Vomiting | 1
  Chest Discomfort | 1
  Device Breakage | 2
  Oropharyngeal Pain | 4
  Throat Irritation | 2

ADVERSE EVENTS:
Time Frame: Subjects will be contacted 7 days (+/- 2 days) following the Cytosponge and upper endoscopy procedures. During this phone call, adverse events will be assessed and subjects will complete questionnaires. Participation in the study is complete when subjects have completed the follow-up phone call.
Groups:
- Patient Wth Barrett's: Subjects presenting for routine endoscopic BE surveillance examinations who had at least a C1 or M3 segment confirmed (or medically suspected).
  Cytosponge™ Cell Collection Device: Cytosponge™ Cell Collection Device is indicated for use in the collection and retrieval of surface cells in the esophagus.
- Patients With GERD: Subjects with gastroesophageal reflux disease (GERD) symptoms undergoing screening for BE
  Cytosponge™ Cell Collection Device: Cytosponge™ Cell Collection Device is indicated for use in the collection and retrieval of surface cells in the esophagus.
Arm/Group | Patient Wth Barrett's | Patients With GERD
All-Cause Mortality (participants affected / at risk) | 0/129 | 0/62
Serious Adverse Events (participants affected / at risk) | 2/129 | 0/62
Other Adverse Events (participants affected / at risk) | 8/129 | 6/62
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Patient Wth Barrett's (N=129) | Patients With GERD (N=62)
Sponge Detachment (Product Issues) | 2 (2) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Patient Wth Barrett's (N=129) | Patients With GERD (N=62)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2)
Throat Irritation (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1)
Device Breakage (Product Issues) | 2 (2) | 0 (0)
Chest Discomfort (General disorders) | 1 (1) | 0 (0)
Not Coded (Investigations) | 2 (2) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2017-12-01): https://cdn.clinicaltrials.gov/large-docs/71/NCT02395471/Prot_000.pdf
  • Statistical Analysis Plan (2018-08-20): https://cdn.clinicaltrials.gov/large-docs/71/NCT02395471/SAP_001.pdf